CLINICAL TRIAL: NCT03699137
Title: Use and Impact of the Pre-hospital 12-lead Electrocardiogram in the Primary PCI Era: Mixed Methods Study (PHECG2)
Brief Title: Pre-hospital ECG in Acute Coronary Syndromes
Acronym: PHECG2
Status: Completed | Type: Observational
Sponsor: Kingston University (Other)
Collaborators: Swansea University (Other); University of Leeds (Other); London Ambulance Service (Other); West Midlands Ambulance Service NHS Foundation Trust (Unknown); South West Ambulance Service NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: ECCCR_PHECG2
Record Dates: First submitted 2018-09-18; First posted 2018-10-09 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Acute Coronary Syndrome; STEMI; Non STEMI
Keywords: Acute coronary syndrome; Emergency Medical Services; Electrocardiogram; Outcomes
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases with confirmed ACS: Cases with confirmed diagnosis of acute coronary syndrome in the MINAP database (national registry of ACS patients). No interventions apply to this group as this is an observational study.
  Interventions: Other: No interventions
- EMS personnel: Emergency Medical Service (EMS) personnel will take part in the focus group. No intervention applies to this group in this qualitative component of the study.
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
The Pre-Hospital 12-lead electrocardiogram (PHECG) is a simple test that helps ambulance clinicians assess patients with suspected acute coronary syndrome (heart attack), and provides clinical data to inform ongoing care. This project builds on previous work by this team, which found that one in three eligible patients did not receive a PHECG, but those that did had a lowered risk of short-term death. In this study the investigators will update that work, and explore reasons for variations in practice - highlighting opportunities to improve care and outcomes.

Using routinely collected data and qualitative methods, the investigators will research patient, practitioner and contextual factors contributing to the decision to administer a PHECG. The aim is also to develop an intervention to increase the proportion of eligible patients that receive a PHECG, and to produce a proposal for further funding to test this intervention in a subsequent randomised trial.

DETAILED DESCRIPTION:
This mixed methods design study consists of four work packages:

WP1 - Population-based, linked cohort study using MINAP data from 2010-2016

This work package will entail analysis of data from around 420,000 pseudonymised patient records from the MINAP database, linking to the Office for National Statistics (ONS) in order to determine mortality/vital status. No patients will be contacted to obtain consent for inclusion of their records in the study as NICOR (custodian of MINAP data) hold section 251 exemption to hold and process patient data for clinical audit purposes without their explicit consent. The data will be released to the research team, using established processes, in pseudonymised format.

The study statisticians will analyse the data provided from MINAP to determine how many heart attack patients who came by ambulance survive to 30 days, estimate time to death, and will estimate from the data whether more people who had an ambulance ECG survive compared to those who did not have the test.

The aim of the study is also to determine from the data whether patients who have an ambulance ECG receive treatment in hospital faster than those who did not.

WP2 - Retrospective chart review of ambulance records

The study statisticians will generate from the larger sample discussed above, a smaller sample (approximately 1800 patients in total) specific to three National Health Service (NHS) ambulance services (Welsh, West Midlands and South West). The investigators will then work with those ambulance services to review the records held by the ambulance service, to see what other information over and above that is collected in the national MINAP audit (e.g. presenting symptoms, severity of any chest pain, public place or home, patient preferences including declining to have the test, ambulance clinician grade and gender). The investigators have worked with a 'task and finish group' of paramedics and cardiology experts to agree which data might be helpful and devised specific forms to collect these data. Data collection from ambulance records will be undertaken by NHS paramedics in the three ambulance services, seconded to work on this project. These paramedics will receive specific training in study procedures to ensure accuracy and data quality. Anonymised data collected by these 'research paramedics' will be sent to the research team by secure electronic database.

WP3 - Ambulance clinician self-report on PHECG recording

In this work package, clinical staff from the three participating ambulance Trusts (48 in total) will be invited to participate in focus group discussions led by an experienced researcher. A semi-structured topic guide (developed beforehand with the help and advice of a small group of paramedics and cardiac experts, and our knowledge of previous literature on paramedic decision making) will be used to explore the view of consenting ambulance clinicians about their perceptions of the role of the PHECG, their experiences of assessing patients with suspected heart attack, and factors which might influence the decision to record (or not) an ECG when assessing and treating a patient.

Focus group discussions will be audio-recorded and transcribed. A method called framework analysis will be used to analyse the transcribed records of the focus group discussions to see whether any particular themes arise, including consensus or disagreement of ambulance staff views on recording an ECG, and consider them against any differences in the characteristics of focus group participants (e.g. grade of clinician, employing ambulance service's local practice).

WP4 - Synthesis of the findings

The investigators will bring together ambulance staff, patient representatives, cardiac experts and researchers to consider the findings from the three work packages described above, with aim to synthesise the study findings and present evidence addressing the study research questions. This will be done with consideration of the investigators' work as forming the 'development phase' for the design of a complex intervention for further testing in a later study.

The project has been designed with input from patient and public representatives especially around the importance of the research question(s), potential impact of the findings for patients and the public. The study team includes three paramedics who have been instrumental in the design of the study as well as supporting documentation particularly for WP3.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Patients with ACS
* Patients who have been brought to hospital by Emergency Medical Service (EMS)
* Patients included in the MINAP registry
* First episode of ACS
* Patients with confirmed STEMI and NSTEMI
* EMS personnel trained in performing an ECG in the pre-hospital setting
* EMS personnel involved in care of patients with a suspected heart attack

Exclusion Criteria:

* patients < 18 years of age
* patients who self-presented at hospitals with suspected ACS
* patients who developed ACS whilst in hospital

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two types of study populations:
  1. - Patients with confirmed diagnosis of ACS in MINAP database as per inclusion and exclusion criteria
  2. - Emergency Medical Service personnel who have been trained to perform 12 lead ECG.
Sampling Method: Non-Probability Sample
Enrollment: 420048 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
WP1: 30-day mortality | 30 days
  Proportion of patients who die within 30 days of the date of their event

SECONDARY OUTCOMES:
Time to death | Up to one year
  Length of time in days from ACS event to death
Hospital mortality | Up to 90 days
  Proportion of patients in each group who die during the (initial) hospital stay following their event
One year mortality | One year
  Proportion of patients in each group who die within one year of their ACS event.
Time under care of EMS | Up to 3 hours
  Length of time from EMS arrival on scene to patient arrives at hospital.
Use and type of reperfusion | 24 hours
  Proportion of patients with STEMI who receive reperfusion treatment (pPCI or fibrinolytic).
Time to treatment | 24 hours
  Time in minutes from initial EMS call to patients first recorded reperfusion treatment.(STEMI only)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Quinn, FESC FAHA FACC, Principal Investigator — Kingston University & St George's, University of London
Locations (3):
- United Kingdom (3):
  - South Western Ambulance Service NHS Foundation Trust, Exeter, Devon
  - Welsh Ambulance Services NHS Trust, Cardiff, Wales
  - West Midlands Ambulance Service, Brierley Hill, West Midlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Welsford M, Nikolaou NI, Beygui F, Bossaert L, Ghaemmaghami C, Nonogi H, O'Connor RE, Pichel DR, Scott T, Walters DL, Woolfrey KG; Acute Coronary Syndrome Chapter Collaborators. Part 5: Acute Coronary Syndromes: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2015 Oct 20;132(16 Suppl 1):S146-76. doi: 10.1161/CIR.0000000000000274. No abstract available. PMID 26472852
- [Background] O'Connor RE, Al Ali AS, Brady WJ, Ghaemmaghami CA, Menon V, Welsford M, Shuster M. Part 9: Acute Coronary Syndromes: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S483-500. doi: 10.1161/CIR.0000000000000263. No abstract available. PMID 26472997
- [Background] Nikolaou NI, Arntz HR, Bellou A, Beygui F, Bossaert LL, Cariou A; Initial management of acute coronary syndromes section Collaborator. European Resuscitation Council Guidelines for Resuscitation 2015 Section 8. Initial management of acute coronary syndromes. Resuscitation. 2015 Oct;95:264-77. doi: 10.1016/j.resuscitation.2015.07.030. Epub 2015 Oct 15. No abstract available. PMID 26477416
- [Background] Tubaro M, Danchin N, Goldstein P, Filippatos G, Hasin Y, Heras M, Jansky P, Norekval TM, Swahn E, Thygesen K, Vrints C, Zahger D, Arntz HR, Bellou A, De La Coussaye JE, De Luca L, Huber K, Lambert Y, Lettino M, Lindahl B, McLean S, Nibbe L, Peacock WF, Price S, Quinn T, Spaulding C, Tatu-Chitoiu G, Van De Werf F. Pre-hospital treatment of STEMI patients. A scientific statement of the Working Group Acute Cardiac Care of the European Society of Cardiology. Acute Card Care. 2011 Jun;13(2):56-67. doi: 10.3109/17482941.2011.581292. PMID 21627394
- [Background] Quinn T, Johnsen S, Gale CP, Snooks H, McLean S, Woollard M, Weston C; Myocardial Ischaemia National Audit Project (MINAP) Steering Group. Effects of prehospital 12-lead ECG on processes of care and mortality in acute coronary syndrome: a linked cohort study from the Myocardial Ischaemia National Audit Project. Heart. 2014 Jun;100(12):944-50. doi: 10.1136/heartjnl-2013-304599. Epub 2014 Apr 14. PMID 24732676
- [Background] Curtis JP, Portnay EL, Wang Y, McNamara RL, Herrin J, Bradley EH, Magid DJ, Blaney ME, Canto JG, Krumholz HM; National Registry of Myocardial Infarction-4. The pre-hospital electrocardiogram and time to reperfusion in patients with acute myocardial infarction, 2000-2002: findings from the National Registry of Myocardial Infarction-4. J Am Coll Cardiol. 2006 Apr 18;47(8):1544-52. doi: 10.1016/j.jacc.2005.10.077. Epub 2006 Mar 29. PMID 16630989
- [Background] Diercks DB, Kontos MC, Chen AY, Pollack CV Jr, Wiviott SD, Rumsfeld JS, Magid DJ, Gibler WB, Cannon CP, Peterson ED, Roe MT. Utilization and impact of pre-hospital electrocardiograms for patients with acute ST-segment elevation myocardial infarction: data from the NCDR (National Cardiovascular Data Registry) ACTION (Acute Coronary Treatment and Intervention Outcomes Network) Registry. J Am Coll Cardiol. 2009 Jan 13;53(2):161-6. doi: 10.1016/j.jacc.2008.09.030. PMID 19130984
- [Background] Ducas RA, Labos C, Allen D, Golian M, Jeyaraman M, Lys J, Mann A, Copstein L, Vokey S, Rabbani R, Zarychanski R, Abou-Setta AM, Menkis AH. Association of Pre-hospital ECG Administration With Clinical Outcomes in ST-Segment Myocardial Infarction: A Systematic Review and Meta-analysis. Can J Cardiol. 2016 Dec;32(12):1531-1541. doi: 10.1016/j.cjca.2016.06.004. Epub 2016 Jun 14. PMID 27707525
- [Background] Surveillance report 2016 - Unstable angina and NSTEMI (2010) NICE guideline CG94 and Myocardial infarction with ST-segment elevation (2013) NICE guideline CG167 [Internet]. London: National Institute for Health and Care Excellence (UK); 2016 Sep 29. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK552026/ PMID 31886964
- [Background] Klerdal K, Varenhorst C, James S, Alfredsson L, Blomberg H, Moradi T. Sex as a determinant of prehospital ECG in ST- and non-ST elevation myocardial infarction patients. Heart. 2014 Nov;100(22):1817-8. doi: 10.1136/heartjnl-2014-306412. Epub 2014 Jul 24. No abstract available. PMID 25060757
- [Background] Coventry LL, Finn J, Bremner AP. Sex differences in symptom presentation in acute myocardial infarction: a systematic review and meta-analysis. Heart Lung. 2011 Nov-Dec;40(6):477-91. doi: 10.1016/j.hrtlng.2011.05.001. PMID 22000678
- [Background] Cioffi J. A study of the use of past experiences in clinical decision making in emergency situations. Int J Nurs Stud. 2001 Oct;38(5):591-9. doi: 10.1016/s0020-7489(00)00096-1. PMID 11524105
- [Background] Croskerry P. Achieving quality in clinical decision making: cognitive strategies and detection of bias. Acad Emerg Med. 2002 Nov;9(11):1184-204. doi: 10.1111/j.1553-2712.2002.tb01574.x. PMID 12414468
- [Background] Hall KH. Reviewing intuitive decision-making and uncertainty: the implications for medical education. Med Educ. 2002 Mar;36(3):216-24. doi: 10.1046/j.1365-2923.2002.01140.x. PMID 11879511
- [Background] Tversky A, Kahneman D. Judgment under Uncertainty: Heuristics and Biases. Science. 1974 Sep 27;185(4157):1124-31. doi: 10.1126/science.185.4157.1124. PMID 17835457
- [Background] Porter A, Snooks H, Youren A, Gaze S, Whitfield R, Rapport F, Woollard M. "Covering our backs": ambulance crews' attitudes towards clinical documentation when emergency (999) patients are not conveyed to hospital. Emerg Med J. 2008 May;25(5):292-5. doi: 10.1136/emj.2007.050443. PMID 18434469
- [Background] Snooks HA, Kearsley N, Dale J, Halter M, Redhead J, Foster J. Gaps between policy, protocols and practice: a qualitative study of the views and practice of emergency ambulance staff concerning the care of patients with non-urgent needs. Qual Saf Health Care. 2005 Aug;14(4):251-7. doi: 10.1136/qshc.2004.012195. PMID 16076788
- [Background] O'Hara R, Johnson M, Siriwardena AN, Weyman A, Turner J, Shaw D, Mortimer P, Newman C, Hirst E, Storey M, Mason S, Quinn T, Shewan J. A qualitative study of systemic influences on paramedic decision making: care transitions and patient safety. J Health Serv Res Policy. 2015 Jan;20(1 Suppl):45-53. doi: 10.1177/1355819614558472. PMID 25472989
- [Background] 19. MRC. Developing and evaluating complex interventions: new guidance. 2006. Accessed at https://www.mrc.ac.uk/documents/pdf/complex-interventions-guidance/ June 2017.
- [Background] Creswell J and Plano Clark V. Designing and conducting mixed methods research. Second Edition 2006; Sage.
- [Background] National Institute for Cardiovascular Outcomes Research. Myocardial Ischaemia National Audit Project. Heart attack in England, Wales and Northern Ireland. Annual Public Report April 2015 - March 2016. June 2017.
- [Background] Kaji AH, Schriger D, Green S. Looking through the retrospectoscope: reducing bias in emergency medicine chart review studies. Ann Emerg Med. 2014 Sep;64(3):292-8. doi: 10.1016/j.annemergmed.2014.03.025. Epub 2014 Apr 18. No abstract available. PMID 24746846
- [Background] McHugh ML. Interrater reliability: the kappa statistic. Biochem Med (Zagreb). 2012;22(3):276-82. PMID 23092060
- [Background] Ritchie J, Lewis J, Nicholls CMN, et al. Qualitative research practice: A guide for social science students and researchers. Sage 2013.
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] National Institute for Health and Clinical Excellence. Behaviour Change at Population, Community and Individual Levels. NICE Public Health Guidance. London: NICE, 2007
- [Background] Heaton J, Day J, Britten N. Collaborative research and the co-production of knowledge for practice: an illustrative case study. Implement Sci. 2016 Feb 20;11:20. doi: 10.1186/s13012-016-0383-9. PMID 26897169
- [Background] Schiele F, Gale CP, Bonnefoy E, Capuano F, Claeys MJ, Danchin N, Fox KA, Huber K, Iakobishvili Z, Lettino M, Quinn T, Rubini Gimenez M, Botker HE, Swahn E, Timmis A, Tubaro M, Vrints C, Walker D, Zahger D, Zeymer U, Bueno H. Quality indicators for acute myocardial infarction: A position paper of the Acute Cardiovascular Care Association. Eur Heart J Acute Cardiovasc Care. 2017 Feb;6(1):34-59. doi: 10.1177/2048872616643053. Epub 2016 Sep 20. PMID 27574334
- [Background] Kvale, S. InterViews: An introduction to qualitative research interviewing. Thousand Oaks, CA: Sage 1996.
- [Background] Ji C, Quinn T, Gavalova L, Lall R, Scomparin C, Horton J, Deakin CD, Pocock H, Smyth MA, Rees N, Brace-McDonnell SJ, Gates S, Perkins GD. Feasibility of data linkage in the PARAMEDIC trial: a cluster randomised trial of mechanical chest compression in out-of-hospital cardiac arrest. BMJ Open. 2018 Jul 28;8(7):e021519. doi: 10.1136/bmjopen-2018-021519. PMID 30056384
- [Derived] Gavalova L, Halter M, Snooks H, Gale CP, Weston C, Watkins A, Munro S, Davies G, Hampton C, Driscoll T, Rosser A, Rees N, Black S, Quinn T. Use and impact of the prehospital 12-lead ECG in the primary PCI era (PHECG2): protocol for a mixed-method study. Open Heart. 2019 Dec 2;6(2):e001156. doi: 10.1136/openhrt-2019-001156. eCollection 2019. PMID 31803487
- See also: What is NVivo — https://www.qsrinternational.com/nvivo-qualitative-data-analysis-software/home